CLINICAL TRIAL: NCT01285973
Title: Evaluation of Integra® Artificial Dermis for the Treatment of Leg Ulcers
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Services (Industry)
Responsible Party: Sponsor
Other Study IDs: RECON-EMEA-10
Record Dates: First submitted 2011-01-27; First posted 2011-01-28 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Lower Limb Ulcer
MeSH Terms: conditions — Leg Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this prospective study is to assess the utility of treatment of leg ulcers using a skin substitute, Integra®, assessing the quality of wound skin healing and transcutaneous oxygen pressure in the distal region of the wound.

This is a multi-centre study on 60 patients who have a lower limb ulcer.

ELIGIBILITY:
Inclusion Criteria:

* patient with a lower limb ulcer, regardless of origin (arterial, venous or mixed, diabetic foot ulcer) present for more than 6 months or large in size (> 10 cm²)
* patients in whom the surgeon has recommended that an Integra® matrix be implanted (even if the patient is not taking part in the study) before the dermo-epidermal graft to obtain a richly vascularised neodermis.
* not eligible for skin flap surgery,
* the patient or patient's representative has agreed to sign the information letter before any investigation required by the research.

Exclusion Criteria:

* circumferential wound,
* wound infection
* immunosuppressed patient,
* known allergy to bovine collagen, bovine glycosaminoglycans or silicone,
* patients under legal guardianship,
* pregnant women
* patients whose health would compromise follow-up for at least 18 months,
* patients whose mental health would compromise completion of the self-evaluation questionnaires.
* wound located in an area not visible by the patient (as no self-assessment would be possible).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients with "difficult" lower limb ulcers, whose wounds have not responded to directed healing for more than 6 months or who have a wound > 10 cm².
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a greater than 50% reduction in wound surface area during the 18 months after grafting. | 18 months

SECONDARY OUTCOMES:
Functional complications of healing at 3, 6, 12 and 18 months | 3, 6, 12 and 18 months
Complete wound healing (reduction in wound surface area >90%) | 3, 6, 12, 18 months
Pain | 3, 6, 12, 18 months
Quality of life | 3, 6, 12, 18 months
Transcutnaeous oxygen pressure (TcPO2) | 6, 12 and 18 months

CONTACTS AND LOCATIONS:
Locations (3):
- Bordeaux University Hospital,, Bordeaux, France
- Aristotle University of Thessaloniki - Papageorgiou General Hospital, Thessaloniki, Greece
- Policlinico Universitario "G. Martino", Messina, Italy